CLINICAL TRIAL: NCT01188759
Title: A Prospective, Randomized Trial Comparing The Safety, Tolerability, And Efficacy Of Voriconazole And Anidulafungin In Combination To That Of Voriconazole Alone When Used For Primary Therapy Of Invasive Aspergillosis in Pediatric Subjects Aged 2 to 17 Years
Brief Title: Voriconazole And Anidulafungin Combination For Invasive Aspergillosis In Pediatric Subjects
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A1501095
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Last update posted 2012-05-11 (Estimated); Status verified 2012-05

CONDITIONS: Aspergillosis; Invasive Pulmonary Aspergillosis; Neuroaspergillosis
Keywords: Aspergillosis; Combination Therapy; Voriconazole; Anidulafungin
MeSH Terms: conditions — Aspergillosis; Invasive Pulmonary Aspergillosis; Neuroaspergillosis | interventions — Voriconazole; Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voriconazole and Anidulafungin Combination (Experimental): Subjects in the combination arm will receive voriconazole and anidulafungin in combination for 2-4 weeks followed by voriconazole monotherapy to complete 6-12 weeks of therapy.
  Interventions: Drug: Voriconazole; Drug: Anidulafungin
- Voriconazole Monotherapy (Active Comparator): Subjects in the monotherapy arm will receive voriconazole monotherapy for 6-12 weeks of therapy.
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — For Children aged 2-11 years and adolescents aged 12-14 years weighing <50 kg:
  Voriconazole 9 mg/kg IV load q12h x 24h, then 8 mg/kg IV q12h, with option to switch to oral voriconazole at 9 mg/kg q12h (maximum 350 mg) after 7 days.
  For adolescents aged 12-17 years, excluding 12-14-year-olds weighing <50kg:
  Voriconazole 6 mg/kg IV q12h x 24h, then 4 mg/kg IV q12h, with an option to switch to oral voriconazole at 200 mg q12h after 7 days.
  Voriconazole therapy is to be given for 6-12 weeks.
  Arms: Voriconazole and Anidulafungin Combination
Drug: Anidulafungin — Anidulafungin 3 mg/kg IV load q24h x 24h (maximum 200 mg), then 1.5 mg/kg q24h (maximum 100 mg).
  Anidulafungin therapy is to be given for 2-4 weeks in combination with voriconazole.
  Arms: Voriconazole and Anidulafungin Combination
Drug: Voriconazole — For Children aged 2-11 years and adolescents aged 12-14 years weighing <50 kg:
  Voriconazole 9 mg/kg IV load q12h x 24h, then 8 mg/kg IV q12h, with option to switch to oral voriconazole at 9 mg/kg q12h (maximum 350 mg) after 7 days.
  For adolescents aged 12-17 years, excluding 12-14-year-olds weighing <50kg:
  Voriconazole 6 mg/kg IV q12h x 24h, then 4 mg/kg IV q12h, with an option to switch to oral voriconazole at 200 mg q12h after 7 days.
  Voriconazole therapy is to be given for 6-12 weeks.
  Arms: Voriconazole Monotherapy

SUMMARY:
This study aims to compare the safety, tolerability, and efficacy of voriconazole and anidulafungin in combination versus voriconazole alone in pediatric subjects aged 2 to 17 years with invasive aspergillosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of proven, probable, or possible invasive aspergillosis.
* Hematologic malignancy or allogeneic hematopoetic stem cell transplant.

Exclusion Criteria:

* Sarcoidosis, aspergilloma, or allergic bronchopulmonary aspergillosis.
* Chronic invasive aspergillosis.
* Receipt of antifungal treatment for more than 96 hours.
* Severe liver dysfunction.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of voriconazole and anidulafungin in combination versus voriconazole alone as determined by rates of adverse events | 12 weeks

SECONDARY OUTCOMES:
Rate of all-cause mortality at 6 weeks | 6 weeks
Rate of all-cause mortality at EOT | 12 weeks
Global response to therapy at 6 weeks | 6 weeks
Global response to therapy at EOT | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501095&StudyName=Voriconazole%20And%20Anidulafungin%20Combination%20For%20Invasive%20Aspergillosis%20In%20Pediatric%20Subjects